CLINICAL TRIAL: NCT02313454
Title: A Single Center, Randomized, Controlled, Single-Masked, Cross-Over Clinical Pilot Study to Evaluate the Reduction in the Exacerbation of the Symptoms of Dry Eye Upon Exposure to a Controlled Adverse Environment (CAESM) With Treatment by the Oculeve Nasal Lacrimal TENS Unit
Brief Title: Evaluation of the Safety and Effectiveness of the Oculeve Intranasal Lacrimal Neurostimulator in Patients With Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OCUN-007
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye syndrome; keratoconjunctivitis; ophthalmic; eye disease; corneal disease; keratitis
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis; Eye Diseases; Corneal Diseases; Keratitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Intranasal Application (Experimental): Intranasal Tear Neurostimulator device, intranasal application for approximately 3 minutes on Day 0 when the participant experienced an Ocular Discomfort Score (ODS) ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
  Interventions: Device: Intranasal Tear Neurostimulator
- Extranasal Application (Sham Comparator): Intranasal Tear Neurostimulator device, extranasal application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
  Interventions: Device: Intranasal Tear Neurostimulator

INTERVENTIONS:
Device: Intranasal Tear Neurostimulator — Neurostimulation applied intranasally and extranasally.

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of the Intranasal Tear Neurostimulator applied intranasally compared with the same device applied extranasally (control) in treating the symptoms of dry eye exacerbated by the Controlled Adverse Environment (CAE) Model.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral dry eyes
* Capable of providing written informed consent

Exclusion Criteria:

* Chronic or recurring epistaxis (nosebleeds)
* Uncontrolled systemic disease
* Blood coagulation disorder
* Females who are pregnant, nursing or planning a pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2015-04-08 (Actual); Study Completion 2015-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Study Chair — Allergan
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were enrolled. 1 participant had an adverse event (pre-existing condition), did not receive treatment and was withdrawn prior to controlled adverse environment (CAE) exposure.
Groups:
- Intranasal Then Extranasal Application: Intranasal Tear Neurostimulator device, intranasal application for approximately 3 minutes at Day 0 when the participant experienced an Ocular Discomfort Score (ODS) ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure; followed by Intranasal Tear Neurostimulator device, extranasal application (control) for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
- Extranasal Then Intranasal Application: Intranasal Tear Neurostimulator device, extranasal application (control) for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure; followed by Intranasal Tear Neurostimulator device, intranasal application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
Period: Treatment 1
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application
Started | 8 (1 participant did not receive the second application.) | 10 (1 participant did not receive the second application.)
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized participants. Intranasal and Extranasal Baseline data are combined because there is only access to combined arm data for this study. The study was acquired from another organization and limited results data are available.
Groups:
- All Participants: Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes at Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure; followed by Intranasal Tear Neurostimulator device, intranasal or extranasal (control) application for approximately 3 minutes on Day 0 when the participant experienced an ODS ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Application to Post-Application in the Ora Calibra Ocular Discomfort Scale (ODS) Score
Description: The participant graded their eye discomfort prior to CAE entry, during CAE exposure to threshold, then starting 1 minute after treatment application every 5 minutes in each eye separately using the Ora Calibra ODS where: 0=no discomfort to 4=constant discomfort. Data from the analysis eye was used to determine effectiveness. The analysis eye was defined as the first eye that reached the threshold and resulted in the device application. If both eyes reached the threshold at the same time point, the analysis eye was the eye with the lowest baseline Schirmer test score (a test to determine if the eye produces enough tears to keep it moist; >10 mm is normal) or, if the Schirmer test scores were equal, the right eye. A negative change from Baseline indicates improvement.
Time Frame: Pre-application to Post-application on Day 0
Population: Per-Protocol (PP) Population was defined as all participants that were able to return to the threshold level following both treatments and did not have any significant protocol violations that might be expected to alter the outcome of their study results.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Extranasal Application: Intranasal Tear Neurostimulator device, extranasal application for approximately 3 minutes on Day 0 when the participant experienced an Ocular Discomfort Score (ODS) ≥3 at 2 or more consecutive time points in at least one eye during CAE exposure.
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 18 | 18
score on a scale | -1.1 (1.0) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Intranasal Application vs Extranasal Application; Test type: Superiority; p = 0.008, Paired t-test; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.0 to -0.19], Standard Deviation 0.8 — Intranasal Application relative to the Extranasal Application

2. Secondary Outcome: Change From Pre-Application to Post-Application in Dry Eye Symptoms (DES) Using a Visual Analog Scale (VAS)
Description: The participant rated their eye dryness (both eyes simultaneously) at all visits and every 5 minutes during CAE exposure by placing a vertical mark on the 100 mm horizontal line to indicate the level of eye dryness. 0 corresponds to "no dryness" and 100 corresponds to "maximal dryness". A negative change from Baseline indicates improvement.
Time Frame: Pre-application to Post-application on Day 0
Population: PP Population was defined as all participants that were able to return to the threshold level following both treatments and did not have any significant protocol violations that might be expected to alter the outcome of their study results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 18 | 18
score on a scale | -18.7 (26.4) | -7.1 (15.9)
Statistical Analysis 1: Comparison: Intranasal Application vs Extranasal Application; Test type: Superiority; p = 0.004, Paired t-test; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-19.0 to -3.4], Standard Error of Mean 15.7 — Intranasal application relative to Extranasal application

ADVERSE EVENTS:
Time Frame: Day 0
Description: Safety Population was defined as all participants from the FAS population.
Arm/Group | Intranasal Application | Extranasal Application
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.